CLINICAL TRIAL: NCT02361996
Title: Quantitative Measurement of Myocardial Perfusion by Cardiac CT in Patients Before and After Coronary-bypass-surgery, Before and After Dilating/Stenting and Before and After Aortic-valve-replacement.
Brief Title: Quantitative Measurement of Myocardial Perfusion by Cardiac CT in Patients
Acronym: CCT/MPERF
Status: Suspended | Type: Observational
Why Stopped: Covid-19 Pandemic
Sponsor: Bakulev Scientific Center of Cardiovascular Surgery (Other Government)
Collaborators: Medical University of Graz (Other); Graz University of Technology (Other)
Responsible Party: Principal Investigator, Rainer Rienmueller, M.D., em.Univ.Prof.Dr.med., Bakulev Scientific Center of Cardiovascular Surgery
Other Study IDs: RENE271242
Record Dates: First submitted 2015-01-15; First posted 2015-02-12 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Coronary Disease; Aortic Valve Stenosis
MeSH Terms: conditions — Coronary Disease; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Coronary Bypass Surgery: inclusion criteria:
  * presence of at least one coronary stenotic lesion above 50% with clinical indication for coronary bypass surgery.
  * list of medication timely related to the procedure
  * signed informed consent
  exclusion criteria:
  * intolerance to contrast agent
  * multiple myeloma, pheochromocytoma, thyroid dysfunction, acute infection
  * renal failure
  * severe arrhythmia
  * pregnancy
  * reduction of cognitive capabilities to understand the purpose and the extent of the study
  * participation in a medical-scientific study using X-rays in the last ten years
  * lack of Russian knowledge to fill the forms
  * lack of signed study agreement
- Coronary Stenting: inclusion criteria:
  * presence of at least one coronary stenotic lesion above 50% with clinical indication for coronary vessel dilatation/stenting.
  * list of medication timely related to the procedure
  * signed informed consent
  exclusion criteria:
  * intolerance to contrast agent
  * multiple myeloma, pheochromocytoma, thyroid dysfunction, acute infection
  * renal failure
  * severe arrhythmia
  * pregnancy
  * reduction of cognitive capabilities to understand the purpose and the extant of the study
  * participation in a medical-scientific study using X-rays in the last ten years
  * lack of Russian knowledge to fill the forms
  * lack of signed study agreement
- Aortic Valve Replacement: inclusion criteria:
  * presence of aortic valve disease (stenosis) with clinical indication for aortic valve replacement without coronary vessel stenosis above 50%
  * list of medication timely related to the procedure
  * signed informed consent
  exclusion criteria:
  * intolerance to contrast agent
  * multiple myeloma, pheochromocytoma, thyroid dysfunction, acute infection
  * renal failure
  * severe arrhythmia
  * pregnancy
  * reduction of cognitive capabilities to understand the purpose and the extent of the study
  * participation in a medical-scientific study using X-rays in the last ten years
  * lack of Russian knowledge to fill the forms
  * lack of signed study agreement

SUMMARY:
It is a common understanding that patients with coronary heart disease are suffering, among others, from reduced myocardial perfusion. In order to increase (normalize) the reduced perfusion, when a conventional approach failed, coronary bypass surgery, coronary vessel dilatation or stenting are performed. The similar situation with reduced myocardial perfusion may be found in patients with stenosis of the aortic valve, where aortic valve replacement may increase myocardial perfusion by left-ventricular remodelling. However, there is presently no method established to measure myocardial perfusion quantitatively and noninvasively before and after a therapeutic intervention.

Data of pre- and post-therapeutic myocardial perfusion, quantitatively measured in ml/100g/min would strengthen the indication for specific therapeutic approach and enable an objective control of effectiveness of the applied therapy.

Hypothesis:

There is a measureable difference in quantitative myocardial perfusion values before (lower) and after (higher) interventional or surgical procedure.

The goal of the study is to measure myocardial perfusion by advanced CT technology (e.g. iCT 256 Brilliance ) quantitatively in ml/100g/min in three groups of patients:

1. Before and after coronary bypass surgery
2. Before and after coronary vessel dilatation/stenting
3. Before and after aortic valve replacement.

The investigators will not assign specific interventions to the subjects of these three groups. Therefore, the research is strictly observational.

Design:

Prospective study to measure quantitatively myocardial perfusion in the above mentioned three groups of patients with simultaneous control and registration of all essential, physiological determinants of myocardial perfusion immediately prior to each CT study. The CT myocardial perfusion measurements will be performed directly after the indication for intervention or surgery and on the last day before discharge from hospital.

All the collected data (determinants) inclusively the CT-studies will be anonymised and archived on a local server. The investigators of the University of Medical Computed Sciences and Technology, Innsbruck / Austria will perform the evaluation of the myocardial perfusion measurements and all statistical analysis independently of the CT-studies performing physicians.

DETAILED DESCRIPTION:
Reliability of the hypothesis:

On phantom studies simulating myocardial perfusion measurements and in animal studies we could confirm that using advanced CT technology (as e.g. "iCT 256 Brilliance") it is possible to measure myocardial perfusion in absolute values - in ml/100g/min. These myocardial perfusion measurements did not differ from those received by EBCT (Electron Beam Computed Tomography). Based on these experimental results and based on the quantitative measurements of myocardial perfusion in 1500 patients studied by EBCT at the Medical University of Graz the hypothesis may be done that using the above mentioned iCT 256 technology, it should be possible to measure myocardial perfusion quantitatively in a daily clinical practice.

Ethical aspects:

The study will be performed according to the international regulations (ISO 14144:212-01) and in agreement with the "Declaration of Helsinki". After oral and written explanation of the planned study and by signing the study agreement by patient and by responsible physician, patients participation is voluntary. The patients participating can leave the study any time without negative sequels for him or her. There is no financial restitution for the patients.

Patients will be informed about (very rare) possible allergoid-toxic reactions during and after intravenous contrast agent application. For possible emergency well trained medical staff and equipment is present. About renal insufficiency: renal failure (creatinin clearance <60ml/min [GFR (Glomerulo Filtration Rate)will be calculated according the Cockroft-Gault-Formula, GFR {ml/min}=((40-age)*weight{kg}*0,85{only for women}]/serum creatinin [mg/dl]*72) above.

The applied X-ray dose (CT) may and will be reduced by:

reduction of KV (kilovoltage) from 120 to 100 or 80 in dependance of patients weight, reduction of MA (milliamper)by using iterative image reconstruction allgorithm (iDOSE). These technical approaches represent the best possibility to reduce X-ray dose for the patient. As the coronary heart disease with stenotic lesions above 50% is a disease mainly of an elderly men (in female mostly after menopause and in male after 50 years of age) the risk for X-Ray dose related genetic defects is very low. The expected applied X-Ray doses by the above mentioned approach will be very low and therefore the risk of X-Ray induced malignancy may be regarded as very low too.

Design:

Prospective study to measure quantitatively myocardial perfusion in the above mentioned three groups of patients with simultaneous control and registration of all essential, physiological determinants of myocardial perfusion immediately before the CT study. The CT myocardial perfusion measurements will be performed directly after the indication for intervention or surgery and on the last day before discharge from hospital.

All the collected data (determinants) including the CT-studies will be anonymised and archived on a local server. These anonymised data may be approached only by members of Graz University of Technology, Institute of Health Care Engineering who will perform the evaluation of the myocardial perfusion measurements and the statistical analysis independently of the CT-studies performing physicians.

Practical procedure:

1. In supine position on CT table the blood pressure and the heart rate will be measured and registered.
2. In all patients a standard native cardiac CT for evaluation of coronary calcification by Agatston score will be performed.
3. In all patients myocardial perfusion will be measured in inspiration and contrast agent application where by the amount of contrast agent and the applied dose is related to patient weights as shown below:

   Patient Perfusion 210mg Iodine/ml Expected dose weight [kg] / [kV/mAs] / [ml] / per shoot [mSv](milli Sievert)

   <60 80/80 40 0.21/ 60-70 80/100 50 0.25/ 70-90 80/120 60 0.30/ 90-100 100/90 70 0.40/ >100 100/100 80 0.43
4. Standard cardiac CT will be performed to evaluate coronary arteries and left ventricular volumes.
5. In supine position on CT table the blood pressure and the heart rate will be measured and registered.

Quantitative evaluation:

The calculation of the myocardial perfusion succeeds in all slices with visible left ventricular myocardium using a modification of the formula described by K.Miles and model based approaches.

The calculation of the left ventricular volumes succeeds by use of the vendors software.

Statistic:

All personal and measured data will be anonymised, tested, analysed and evaluated in Graz University of Technology.

The numerical values will be expressed as mean +/- SD (min, max, 95% CI). p-values of 0.05 will be regarded statistically significant. Paired test and or Wilcoxon signed-rank tests will be used. X² analyses will be used to compare categoric variables. Additionally correlation analyses (Pearson, Spearman) will be performed and method of classification (pre- vs. postoperative) will be applied. All calculation will be done by SPSS 21.0 (SPSS, Chicago, Il, USA) or by Matlab statistic toolbox or R.

The neccessary number of studied patients is based on the results of 64 patients studied before and after aortic valve replacement in whom the myocardial perfusion was measured before and four months after surgery.

Pre-operative: Mean=74 (SD=21) ml/100g/min Post 4 Months: Mean=78 (SD=20) ml/100g/min. Difference= +4ml/100g/min. With 0.5 supposed correlation of the measured values the standard deviation of the differences may be estimated as 20ml/100g/min.

By alpha=0.05, 1-beta=0.80, n=209 patients is needed.

In addition to the pre- and post surgery evaluation, statistical models explaining the influence of collected data on the quantitaitve myocardial perfusion will be computed.

As a drop-out quote of 10% may be expected it is neccessary to study in each group of patients 230 patients. This means total 690 patients.

All data will be registered in database and tested for plausibility.

ELIGIBILITY:
Inclusion Criteria:

in cohort: Coronary Bypass Surgery:

o presence of at least one coronary stenotic lesion above 50% with clinical indication for coronary bypass surgery

in cohort: Coronary Stenting: o presence of at least one coronary stenotic lesion above 50% with indication for coronary vessel dilatation/stenting

in cohort: Aortic Valve Replacement

o presence of aortic valve disease (stenosis) with clinical indication for aortic valve replacement without coronary vessel stenosis above 50%

for all three cohorts:

* list of medication timely related to the procedure
* signed informed consent

Exclusion Criteria:

for all three cohorts:

* intolerance to contrast agent
* multiple myeloma, pheochromocytoma, thyroid dysfunction, acute infection
* renal failure
* severe arrhythmia
* pregnancy
* reduction of cognitive capabilities to understand the purpose and the extent of the study
* participation in a medical-scientific study using X-rays in the last ten years
* lack of Russian knowledge to fill the forms
* lack of signed study agreement -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients above 18 years of age, who are reffered with suspected or known coronary artery disease or aortic valve stenosis either to the Bakoulev Scientific Centre for Cardiovascular Surgery, Moscow / Russia or to the Republican Special Centre of Surgery, Tashkent / Uzbekistan and fulfill the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 690 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change of myocardial perfusion (ml/100g/min) [MPerf] | 2015 - 2019
  after indication for and before intervention or surgery and after intervention or surgery one day before discharge

SECONDARY OUTCOMES:
Composition of parameters influencing the complexity of myocardial perfusion regulation: Heart-rate, blood-pressure, rate-pressure-product, left ventricular haemodynamic parameters | 2015 - 2019
  after indication for and before intervention or surgery and after intervention or surgery one day before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Rainer K Rienmueller, MD, Study Director — Bakoulev Scientific Centre for Cardiovascular Surgery; Medical University Graz; Vladimir N Makarenko, MD, Principal Investigator — Bakoulev Scientific Centre for Cardiovascular Surgery, Moscow / Russia; Marat Khodjibekov, MD, Principal Investigator — Republican Special Center of Surgery, Tashkent / Uzbekistan; Theresa Rienmüller, Dr.techn., Principal Investigator — Graz University of Technology
Locations (3):
- Graz University of Technology, Graz, Austria
- Bakoulev Scientific Center for Cardiovascular Surgery, Moscow, Russia
- Republican Specialized Center of Surgery, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Rienmuller T, Baumgartner C, Handler M, Makarenko V, Ourednicek P, Krestinich IM, Zhorzholiani ST, Rienmuller R, Bockeria L. Quantitative Estimation of Left Ventricular Myocardial Perfusion Based on Dynamic CT Scans. Biomed Tech (Berl). 2013 Aug;58 Suppl 1:/j/bmte.2013.58.issue-s1-L/bmt-2013-4288/bmt-2013-4288.xml. doi: 10.1515/bmt-2013-4288. Epub 2013 Sep 7. No abstract available. PMID 24042936
- [Derived] Lara-Hernandez A, Rienmuller T, Juarez I, Perez M, Reyna F, Baumgartner D, Makarenko VN, Bockeria OL, Maksudov M, Rienmuller R, Baumgartner C. Deep Learning-Based Image Registration in Dynamic Myocardial Perfusion CT Imaging. IEEE Trans Med Imaging. 2023 Mar;42(3):684-696. doi: 10.1109/TMI.2022.3214380. Epub 2023 Mar 2. PMID 36227828
- See also: Bakoulev Scientific Center's Site — https://bakulev.com/
- See also: Site of Graz University of Technology — https://www.tugraz.at/en/institutes/hce/home/